CLINICAL TRIAL: NCT01968746
Title: The AVERT Sepsis Investigation: Assessment of Variability in Early Resuscitation and Treatment of Sepsis
Brief Title: The AVERT Sepsis Investigation
Acronym: AVERT
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Therapeutic Monitoring Systems (Other); MaRS Discovery District (Other)
Responsible Party: Sponsor
Other Study IDs: 602039
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Sepsis; Severe Sepsis
Keywords: Sepsis; Shock
MeSH Terms: conditions — Sepsis; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED patients with suspected infection

SUMMARY:
The overall objective of this study is to utilize heart rate variability and respiratory rate variability in patients with sepsis to predict clinical deterioration and death.

Our specific objectives are:

1. To study the ability of a change in composite variability (∆CVI) assessment to act as a prognostic aid in predicting disease progression in sepsis.
2. To study the effect that standard resuscitation interventions will have on the direction and magnitude of ∆CVI in patients with sepsis.

B. Hypotheses H1: In the initial resuscitation of sepsis, a low or declining multi-parameter composite variability index (CVI) over 4 hours will predict a significant increase in the combined outcome of overt shock, organ dysfunction, and mortality.

H2: In the initial resuscitation of sepsis, low volume fluid resuscitation (<20 cc/kg) over 4 hours will be associated with a low or declining CVI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Antibiotics ordered or administered (as surrogate for suspected or confirmed infection as primary reason for hospital admission as determined by the primary team) 2. Serum lactate ≥ 2.0 mmol/L or transient hypotension (any systolic blood pressure < 100 mmHg).

  3. Identification within 12 hours of a qualifying lactate measurement or hypotension episode 4. Hospital admission planned for suspected infection as primary reasons for admission (per emergency medicine team).

Exclusion Criteria:

* 1. Age < 18 years 2. Pregnancy 3. Non-sinus cardiac rhythm (atrial fibrillation, active pacemaker, SVT) 4. Evidence of Overt Shock upon enrollment:

  * Hypotension: SBP < 90 mmHg for ≥ 60 minutes
  * Any vasopressor or inotrope use (e.g. norepinephrine, dopamine, vasopressin, dobutamine) 5. Acute respiratory support (BiPAP or mechanical ventilation) before enrollment 6. Inability to obtain written informed consent from patient or legally authorized representative 7. Inability to wear Zephyr Bioharness device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted through the ED for suspected infection as primary reason for admission.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progressive organ failure | 72 hours
  A. SOFA score increase by ≥ 1 from baseline B. Overt shock C. Mortality (all-cause, in-hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Arnold, MD, Principal Investigator — Christiana Care Health Services; Andrew JE Seely, MD, PhD, Study Chair — Ottawa Hospital
Locations (5):
- United States (4):
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Health System, Newark, Delaware
  - Billings Clinic, Billings, Montana
  - Cooper University Hospital, Camden, New Jersey
- The Ottawa Hospital, Ottawa, Ontario, Canada